CLINICAL TRIAL: NCT04001595
Title: Global Fukutin-Related Protein Registry
Brief Title: Global FKRP Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Collaborators: LGMD2i Research Fund (Unknown); CureLGMD2i (Unknown); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 23NE0222
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: LGMD2I; LGMDR9; Limb Girdle Muscular Dystrophy; Congenital Muscular Dystrophy; Muscle-Eye-Brain Disease; Walker-Warburg Syndrome; FKRP Gene Mutation
Keywords: LGMD2I; LGMDR9; Limb Girdle Muscular Dystrophy; Congenital Muscular Dystrophy; Muscle-Eye-Brain Disease; Walker-Warburg Syndrome; FKRP gene mutation
MeSH Terms: conditions — Muscular Dystrophy, Limb-Girdle, Type 2I; Muscular Dystrophies, Limb-Girdle; Walker-Warburg Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with FKRP gene mutation
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — Participants who have volunteered to participate will complete various questionnaires relating to their condition.

SUMMARY:
Mutations in the Fukutin Related Protein (FKRP) gene cause the condition Limb Girdle Muscular Dystrophy type R9 (LGMDR9) also known as LGMD2I, and the rarer conditions Congenital Muscular Dystrophy (MDC1C), Muscle Eye Brain Disease (MEB) and Walker-Warburg Syndrome (WWS). LGMDR9 is the most common FKRP-related condition, and is especially prevalent in Northern Europe.

The aim is to facilitate a questionnaire based research study in order to better characterise and understand the disease globally. By maintaining a global registry this will help identify potential participants eligible for clinical trials in the future.

DETAILED DESCRIPTION:
The Global FKRP Registry (https://www.fkrp-registry.org/) is an international registry for patients with an FKRP-related condition; no experimental intervention is involved. Patients will receive information on the most up to date standards of care relating to their disease and may be invited to participate in relevant clinical trials. Their data will be updated annually and stored indefinitely, or until they request their data to be removed.

The data will be collected via an online form and will be stored on a secure server based in the United Kingdom and looked after by the registry staff at Newcastle University. Data collected from patients will include demographic information, diagnosis, current condition, age of onset, medication, contractures, family history and results of genetic testing, if available. Other optional questionnaires will focus on patients' pain and quality of life. Further information collected from patients' doctors will include, heart and lung function, muscle strength, muscle and brain MRI findings and genetics.

The FKRP registry is funded by LGMD2i Research Fund and CureLGMD2i.

The primary objectives of the Global FKRP Registry are to:

* Accelerate and facilitate clinical trials by locating potential research subjects quickly and efficiently
* Facilitate in the planning of clinical trials
* Assist the neuromuscular community with the development of recommendations and standards of care
* Characterise and describe the FKRP population as a whole, enhancing the understanding of the prevalence throughout the world.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a confirmed diagnosis of an FKRP-related condition are eligible for inclusion. Diagnosis will be confirmed via genetic testing results.

Exclusion Criteria:

* There is no exclusion criteria for registration with this patient registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have undergone genetic testing for an FKRP-related condition or have a confirmed diagnosis of an FKRP-related condition can self-register to participate in this study. The study will be advertised through neuromuscular disease clinics, the registry website, patient organisations and conferences.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | 12 months
  Patient-reported FKRP clinical diagnosis, symptoms relating to muscle weakness, motor function and family history.
McGill Pain Questionnaire | 12 months
  Patient-reported current pain.
Individualized Neuromuscular Quality of Life questionnaire (INQoL) | 12 months
  Patient-reported quality of life.
Clinician questionnaire | 12 months
  Doctor-reported clinical data, including respiratory and cardiac test results and genetic confirmation of FKRP mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Straub, MD, PhD, Principal Investigator — John Walton Muscular Dystrophy Research Centre
Locations (1):
- John Walton Muscular Dystrophy Research Centre, Newcastle University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy LB, Schreiber-Katz O, Rafferty K, Robertson A, Topf A, Willis TA, Heidemann M, Thiele S, Bindoff L, Laurent JP, Lochmuller H, Mathews K, Mitchell C, Stevenson JH, Vissing J, Woods L, Walter MC, Straub V. Global FKRP Registry: observations in more than 300 patients with Limb Girdle Muscular Dystrophy R9. Ann Clin Transl Neurol. 2020 May;7(5):757-766. doi: 10.1002/acn3.51042. Epub 2020 Apr 28. PMID 32342672
- [Background] Richardson M, Mayhew A, Muni-Lofra R, Murphy LB, Straub V. Prevalence of Pain within Limb Girdle Muscular Dystrophy R9 and Implications for Other Degenerative Diseases. J Clin Med. 2021 Nov 25;10(23):5517. doi: 10.3390/jcm10235517. PMID 34884219
- See also: Global FKRP Registry website — https://www.fkrp-registry.org/